CLINICAL TRIAL: NCT01099735
Title: Effect of Continuous Positive Airway Pressure On Lower Esophageal Sphincter Pressure in Subjects Undergoing Bariatric Surgery
Brief Title: Effect of Continuous Positive Airway Pressure (CPAP) on Lower Esophageal Sphincter Pressure in Morbidly Obese Patients
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Akram Khan, Principal Investigator, Oregon Health and Science University
Other Study IDs: IRB00005565
Record Dates: First submitted 2010-01-14; First posted 2010-04-07 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Sleep Apnea; Gastroesophageal Reflux Disease
Keywords: Bariatric Surgery; Sleep Apnea; Gastroesophageal Reflux Disease; GERD
MeSH Terms: conditions — Sleep Apnea Syndromes; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CPAP, Manometry: Patients undergoing Manometry before weight loss surgery

SUMMARY:
This trial is enrolling patients who are already being seen at OHSU weight loss clinic or have been referred for clinical reasons by their physician to the OHSU weight loss clinic and are going to have a esophageal manometry that would be paid for by their insurance company for clinical reasons.

In patients undergoing weight loss surgery investigators plan to study the effect of continuous positive airway pressure during a esophageal manometry.

DETAILED DESCRIPTION:
Subjects will be invited to be in this research study because they are being considered for weight loss (bariatric) surgery that is being paid for by their insurance company. As part of the preparation for surgery, subjects will have a test called manometry that measures pressure in the esophagus (food pipe). For this test, a tube will be lowered down one nostril into the food pipe.

Studies have shown that Continuous Positive Airway Pressure (CPAP) reduces reflux in people with or without sleep apnea as well as in people with reflux. The investigators are trying to understand how this occurs. This research study will add about 10 additional minutes to the clinic visit. The investigators expect about 50 subjects to be in the study at OHSU. Outcomes will be measured at 18 months.

Patients scheduled for esophageal manometry and motility studies prior to their bariatric surgery will be given a study flyer at the bariatric clinic. A list of the patients who are interested in participating in the study will be given to one of the study investigators. A study investigator will call these patients to explain the study, assess their interest in participation, and review their eligibility for entrance into the study. Assessment of eligibility will be done by asking for medical history over the phone as well as by requesting access to their medical record to ensure the patients do not meet exclusion criteria. After review of the patient's clinical history verbally and through review of the medical record, informed consent will be signed at their manometry appointment.

Subjects will undergo the manometry procedure. After finishing the procedure, when the catheter would normally be withdrawn after the procedure, it will remain in place for the study. A CPAP mask will be placed over the subject's nose. CPAP blows air in the nose with a mild pressure. The air pressure will be slowly increased while pressure in the esophagus is being recorded. As done with the regular manometry, the subject will be asked to swallow small amounts of water during the test. The test will be completed in 10 minutes. The CPAP and the tube will be removed.

Subjects will complete a questionnaire prior to the manometry about gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria

1. Adult > 18 yrs old
2. Willing to give informed consent
3. Undergoing bariatric surgery and scheduled to undergo manometry and polysomnography as part of the protocol.

Exclusion Criteria

1. Patient unwilling to give informed consent
2. Pregnant women
3. Patients with prior history of esophageal surgery (e.g. Nissen fundoplication, partial resection, dilation, stent placement), known anatomic abnormality of the esophagus (e.g. stricture, Schatzki's ring, Zenker's diverticulum, malignancy, varices, ulcers), and/or known functional abnormality of the esophagus (e.g. achalasia, dysmotility).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Lower Esophageal Sphincter Pressure | 18 months
  Effect of CPAP on Lower esophageal sphincter pressure will be assessed after 18 months of data collection or after all 50 patients have been assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- See also: OHSU Pulmonary Critical Care Medicine — http://www.ohsu.edu/pccm/